CLINICAL TRIAL: NCT00971009
Title: Effects of Internet Support for Cancer Patients on Health Outcomes, Health Care Utilization and Costs: A Randomized Clinical Trial
Brief Title: Effects of Internet Support for Cancer Patients
Acronym: WebChoice 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Cornelia Ruland, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009051
Record Dates: First submitted 2009-09-01; First posted 2009-09-03 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Symptom management; Interactive Health Communication Application; Patient-provider communication; Health care costs
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- OPPC service (Experimental): A practice-integrated nurse administered online patient-provider communication (OPPC) service including access to asking questions to social counselors
  Interventions: Behavioral: OPPC service
- WebChoice IHCA (Experimental): WebChoice is an interactive health communications application (IHCA) that in addition to offer a practice-integrated nurse administered online patient-provider communication (OPPC) service, allows patients to monitor their symptoms and health problems from home; provides them with individually tailored, just-in-time information and support to manage their symptoms and illness-related problems between treatments and during rehabilitation; and a forum, or e-group community, for group discussion with other cancer patients.
  Interventions: Behavioral: WebChoice IHCA
- Control group (No Intervention): The control group receives usual care

INTERVENTIONS:
Behavioral: OPPC service — Access to a practice-integrated nurse administered online patient-provider communication (OPPC) service including access to asking questions to social counselors
  Arms: OPPC service
Behavioral: WebChoice IHCA — The additional features of WebChoice allows patients to monitor their symptoms and health problems from home; provides them with individually tailored, just-in-time information and support to manage their symptoms and illness-related problems between treatments and during rehabilitation; and a forum, or e-group community, for group discussion with other cancer patients.
  Arms: WebChoice IHCA

SUMMARY:
Being diagnosed and treated for cancer is usually associated with severe physical symptoms, impaired functional status, complex emotional, psychosocial and existential issues and substantial worries. Failure to help patients with their problems and worries can unnecessarily delay patients' recovery and rehabilitation, lead to chronic functional impairments, anxiety and depression and prolong patients' needs for health care and social services. The objectives of this interdisciplinary, international research project that includes collaboration with HELFO (The Norwegian Health Economy Administration), are to test and compare, in a randomized, controlled trial (RCT), the effects of (1) a practice-integrated online patient-provider communication (OPPC) service including access to asking questions to HELFO, (2) a multi-component Interactive Health Communication Application (IHCA) called WebChoice, and (3) usual care on: patient outcomes, health care and social services use and costs. Breast cancer patients undergoing treatment at three different hospitals in Norway will be randomized into two experimental and one control groups and will be followed with 5 repeated measures over one year. The proposed study will contribute to innovative methods and technologies that can radically improve patient-provider communication, care quality, and continuity of care. The two interventions tested in this study, the OPPC service with and without additional features of WebChoice, represent new forms of interactions and information sharing between patients and clinicians where patients can get seamless access to communication and information services from where and whenever they need it. This could significantly contribute to reducing unnecessary suffering, less fragmented health care, better efficiency, patient safety, patient satisfaction and have an impact on patients' health services utilization. The investigators' work addresses, therefore, important health policy goals with the potential for considerable societal gains.

ELIGIBILITY:
Inclusion Criteria:

* Patients recently diagnosed with breast cancer and under treatment (radiation, chemotherapy, hormone, or combinations of those)
* Patients are > 18 years of age, able to write / read / speak Norwegian and have Internet with secure access (BankID) at home

Exclusion Criteria:

* Excluded are patients who had received radiation on the brain as this may affect their abilities to reliably report their symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Severity and duration of symptom distress | At baseline and at 2, 4, 6, 8 and 12 months
Anxiety and depression | At baseline an at 2, 4, 6, 8 and 12 months

SECONDARY OUTCOMES:
Self-efficacy | At baseline and at 2, 4, 6, 8 and 12 months
Uncertainty in illness | At baseline and at 2, 4, 6, 8 and 12 months
Health care costs | Post intervention, at 12 and 18 months
Quality of life | At baseline and at 4, 8 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia M Ruland, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital - Rikshospitalet, Oslo, Norway

REFERENCES:
- [Result] Borosund E, Cvancarova M, Moore SM, Ekstedt M, Ruland CM. Comparing effects in regular practice of e-communication and Web-based self-management support among breast cancer patients: preliminary results from a randomized controlled trial. J Med Internet Res. 2014 Dec 18;16(12):e295. doi: 10.2196/jmir.3348. PMID 25525672